CLINICAL TRIAL: NCT02094274
Title: A Single-dose, Randomised, Crossover, Placebo-controlled, Double-dummy, Pharmacodynamic Clinical Trial Assessing Two Fixed Dose Combinations of Long-acting Beta-agonist (LABA) and Inhaled Corticosteroid (ICS)
Brief Title: A Single-dose, Randomised, Crossover, Placebo-controlled Study Assessing Two Fixed-dose Combinations of Inhaled Long-acting Beta-agonist and Corticosteroid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-40468-10; 2013-002939-25 (EudraCT Number)
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAS40468 (Experimental): Single dose, administered via Genuair® dry powder inhaler (DPI)
  Interventions: Drug: LAS40468
- Salmeterol/fluticasone propionate (Active Comparator): Single dose, Seretide® (salmeterol fluticasone propionate) administered via Accuhaler™
  Interventions: Drug: Salmeterol/fluticasone propionate
- Placebo (Placebo Comparator): Single dose administered via Genuair® or Accuhaler™ dry powder inhaler (DPI)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LAS40468
  Arms: LAS40468
Drug: Salmeterol/fluticasone propionate
  Other Names: Seretide®
  Arms: Salmeterol/fluticasone propionate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the the ability of a single dose of LAS40468 administered via Genuair® and a single dose of salmeterol/fluticasone propionate (Seretide®) administered via Accuhaler to produce bronchodilation (opening of the airways) and the safety and tolerability of the treatments

DETAILED DESCRIPTION:
This is a Phase 1, randomised, double-blind, double-dummy, cross-over trial to assess the bronchodilation effect of a single dose of LAS40468 and a single dose of salmeterol/fluticasone propionate (Seretide®) administered to adult patients with stable asthma.

The study will consist of a screening visit and treatment periods of approximately 13 hours separated by washout periods of 7 to 14 days from the time of Investigational Medicinal product (IMP) administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant, non-lactating females aged between 18 and 60 years (both inclusive)
* Patients with a confirmed 6-months' history of asthma at the time of enrolment into the trial
* Patients treated with short-acting beta-agonists or inhaled corticosteroids at a stable dose and regimen (up to the equivalent of 1600 μg/day of beclometasone dipropionate) for at least 4 weeks prior to screening
* Patients whose (pre-salbutamol) forced expiratory volume in 1 second (FEV1) at screening is >60% of the predicted normal value after a washout of at least 6 hours for short-acting beta-agonists and 48 hours for long-acting beta-agonists, if applicable
* Patients with a FEV1 absolute increase of at least 250 mL over baseline value after inhalation of 4 puffs of 100 μg of salbutamol in one of two pulmonary function tests performed within 10-15 min

Exclusion Criteria:

* Patients with clinically significant respiratory or pulmonary diseases other than asthma or history of thoracic surgery
* Patients with a Body Mass Index (BMI) < 18 or > 40kg/m2 (both inclusive)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline (pre-dose at each period) in normalised forced expiratory volume in 1 second (FEV1) area under the curve (AUC) over the 12 hour period after IMP administration (AUC0-12) | 12 Hours

SECONDARY OUTCOMES:
Adverse events | 7-9 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical trial subject (regardless of the administration of the IMP and the causal relationship to it). An AE can therefore be any unfavourable and unintended medical occurrence during subject's participation in the trial, including deterioration of a pre-existing medical, an ECG abnormality, a blood pressure abnormal value or an abnormal finding in the physical examination.
  A Serious AE is any AE that: results in death, is life-threatening, requires hospitalisation or prolongs existing hospitalisation, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is any other medically important event that may jeopardise the subject or may require intervention to prevent one of the other above outcomes. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious AE.

CONTACTS AND LOCATIONS:
Locations (2):
- Almirall Investigational Site #1, Berlin, Germany
- Almirall Investigational Site #2, Harrow, United Kingdom